CLINICAL TRIAL: NCT03749005
Title: Impact of Three-dimensional Visualization on Operation Strategy and Complications for Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201801
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-04

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Three-dimensional Visualization
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the multi-centre study is to evaluate correctly the impact of three dimensional visualization on operation strategy and complications for Pancreatic Cancer.

DETAILED DESCRIPTION:
Because of the complexity of Pancreatic Cancer, the limitations of 2D images of CT/MRI and the uncertainty of surgeons'experience, it is difficult for the surgeons to diagnosis and assess the operation strategy accurately based on traditional 2D imaging(CT/MRI).The aim of the multi-centre study is to evaluate correctly the impact of three-dimensional visualization on operation strategy and complications for Pancreatic Cancer.

ELIGIBILITY:
Inclusion Criteria:

1.18 years≤ Age ≤70 years 2.Compling with the diagnosis criteria of Pancreatic Cancer. 3.Primary Pancreatic Cancer without metastasis. 4.The patients are volunteered for the study.

Exclusion Criteria:

1. Patients with mental illness.
2. Patients can't tolerate the operation owe to a variety of basic diseases (such as severe cardiopulmonary insufficiency, renal insufficiency, cachexia and blood system diseases, etc.)
3. The patients refused to take part in the study.
4. There are other co-existed malignant tumors.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients with Pancreatic Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Impact on operation strategy of three dimensional visualization technique | 30 days
  Firstly, the operation strategies based on original CT or MRI image data will be made by the team, Secondly, the operation strategies based on three dimensional reconstruction models will be made by the team, then, actually surgical strategies will be recorded. The change of operation strategy will be assessed by comparing the strategy of the 2D model and 3D model. The change rate of operation strategy will be recorded and presented as percentage.

SECONDARY OUTCOMES:
Impact on complication of three dimensional visualization technique | 30 days
  The early postoperative complication and mortality are defined as the event observed within 30 days after surgerypostoperative bleeding, biliary fistula, ascites, postoperative liver failure, renal dysfunction, pleural effusion, abdominal cavity infection, abdominal abscess, incision infection, the occurrence cases of each complication (number) will be recorded.
1-year disease free survival rate | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of The Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wu X, Wang D, Xiang N, Pan M, Jia F, Yang J, Fang C. Augmented reality-assisted navigation system contributes to better intraoperative and short-time outcomes of laparoscopic pancreaticoduodenectomy: a retrospective cohort study. Int J Surg. 2023 Sep 1;109(9):2598-2607. doi: 10.1097/JS9.0000000000000536. PMID 37338535
- [Derived] Tao H, Zeng X, Lin W, Wang Z, Lin J, Li J, Qian Y, Yang J, Fang C. Indocyanine green fluorescence imaging to localize insulinoma and provide three-dimensional demarcation for laparoscopic enucleation: a retrospective single-arm cohort study. Int J Surg. 2023 Apr 1;109(4):821-828. doi: 10.1097/JS9.0000000000000319. PMID 37026828